CLINICAL TRIAL: NCT07359924
Title: Application of Liquid Fraction of Platelet-rich Fibrin in Face Care Cream.
Brief Title: PRF in Face Care Cream.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: PUMS-308/18
Record Dates: First submitted 2026-01-13; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Skin Ageing
Keywords: PRF; skin; cream; EGF

STUDY DESIGN:
Intervention Model Description: Patients received three uniformly appearing creams with instruc-tions for application on specific facial areas every morning and evening. Skin reassessment was conducted after 1, 2, and 4 weeks from the start of application. During the four weeks of the study, baseline measurements (elasticity, hydration and transepidermal water loss) were taken weekly, with skin topography and mac-rosculpture additionally examined in weeks 0 and 4.
Who Masked: Participant
Masking Description: Every patients have got identically looking boxes with different creams formulation, signed by following numbers and the instruction for specific application. Every patient received the same instruction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Formulation 1 (Placebo Comparator): Base formulation
  Interventions: Combination Product: The cream base formulation containing oil phase, Creagel EZ® 7 and Alphaflow® 20
- Formulation 2 (Active Comparator): Formulation with growth factor EGF
  Interventions: Combination Product: The cream base formulation containing oil phase, Creagel EZ® 7 and Alphaflow® 20 with additional growth factor EGF
- Formulation 3 (Experimental): Formulation with PRF
  Interventions: Biological: The cream base formulation containing oil phase, Creagel EZ® 7 and Alphaflow® 20 with autologus PRF

INTERVENTIONS:
Combination Product: The cream base formulation containing oil phase, Creagel EZ® 7 and Alphaflow® 20 — Daily skin application for the following 4 weeks at the same place according to the instruction
  Arms: Formulation 1
Combination Product: The cream base formulation containing oil phase, Creagel EZ® 7 and Alphaflow® 20 with additional growth factor EGF — Daily skin application for the following 4 weeks at the same place according to the instruction
  Arms: Formulation 2
Biological: The cream base formulation containing oil phase, Creagel EZ® 7 and Alphaflow® 20 with autologus PRF — Daily skin application for the following 4 weeks at the same place according to the instruction
  Arms: Formulation 3

SUMMARY:
The study evaluates the effectiveness of cosmetic preparations containing PRF, conducted through in vivo studies. Material and Methods: The study involved 20 healthy volunteers (aged 20-40) who received three identically packaged creams to be applied to specific facial areas. Formulation 1: base formulation (control), Formulation 2: base formulation with human epidermal growth factor (EGF), and Formulation 3: base formulation with platelet-rich fibrin (PRF). Volunteers applied the creams as directed for a period of four weeks. Skin assessments was conducted at baseline (week 0), and at weeks 1, 2, and 4. Trans-epidermal Water Loss (TEWL), skin hydration using corneometry to determine the moisture content of the stratum corneum, skin elasticity using a cutometer to measure the skin's ability to return to its original state after deformation, and dermal bioavailability were measured. EGF concentration in the stratum corneum will be measured using the tape-stripping method followed by HPLC (High-Performance Liquid Chroma-tography) analysis. Results: A significant decrease in TEWL was observed in formulations 2 and 3, indicating improved skin barrier function. Formulation 3 showed the highest increase in skin hy-dration, followed by formulation 2. Both formulations 2 and 3 demonstrated improvements in skin elasticity, with formulation 3 showing the greatest enhancement. EGF concentration in the stratum corneum increased over the four-week period, reaching equilibrium with the product concentration by week four. Con-clusion: The in vivo instrumental compatibility studies confirmed that the new cosmetic formulations containing EGF and PRF are safe and effective for human skin.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers with healthy skin, who sign an agreement for study participation

Exclusion Criteria:

* systemic diseases, smoking, blood disorders, acute viral infections and skin inflammations, pregnancy, and breastfeeding.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-02-03 (Actual); Primary Completion 2022-08-08 (Actual); Study Completion 2023-02-06 (Actual)

PRIMARY OUTCOMES:
Skin water content | Baseline
  To measure the hydration of skin, an apparatus called a corneometer is used (Corneometer® CM 825 (Courage+Khazaka electronic GmbH)). It allows an accurate, reproducible and objective measurement of the hydration level of the stratum corneum of the skin. It records changes in electrical capacitance, consistent with the water content of the skin.
Transepidermal water loss | Baseline
  Tewameter
Skin topography | Baseline
  Visioscan® VC98 and Visioline® VL650
Skin elasticity | Baseline
  Cutometer
Dermal Bioavailability | Baseline
  Tape-Stripping Method
Skin water content | After 1 week
  To measure the hydration of skin, an apparatus called a corneometer is used (Corneometer® CM 825 (Courage+Khazaka electronic GmbH)). It allows an accurate, reproducible and objective measurement of the hydration level of the stratum corneum of the skin. It records changes in electrical capacitance, consistent with the water content of the skin.
Skin water content | After 2 weeks
  To measure the hydration of skin, an apparatus called a corneometer is used (Corneometer® CM 825 (Courage+Khazaka electronic GmbH)). It allows an accurate, reproducible and objective measurement of the hydration level of the stratum corneum of the skin. It records changes in electrical capacitance, consistent with the water content of the skin.
Skin water content | After 4 weeks
  To measure the hydration of skin, an apparatus called a corneometer is used (Corneometer® CM 825 (Courage+Khazaka electronic GmbH)). It allows an accurate, reproducible and objective measurement of the hydration level of the stratum corneum of the skin. It records changes in electrical capacitance, consistent with the water content of the skin.
Transepidermal water loss | After 1 week
  Tewameter
Transepidermal water loss | After 2 weeks
  Tewameter
Transepidermal water loss | After 4 weeks
  Tewameter
Skin topography | After 4 weeks
  Visioscan® VC98 and Visioline® VL650
Skin elasticity | After 4 weeks
  Cutometer
Dermal Bioavailability | After 4 weeks
  Tape-Stripping Method

SECONDARY OUTCOMES:
Stability Evaluation of cream formulations | Baseline
  The stability tests of the formulations were carried out immediately after preparation and after 60 days of storage at 40°C. From the obtained results, the arithmetic mean, and standard deviation were calculated. Each sample was tested three times, and the arithmetic mean, and standard deviation were computed from the results.
Stability Evaluation of cream formulations | After 60 days
  The stability tests of the formulations were carried out immediately after preparation and after 60 days of storage at 40°C. From the obtained results, the arithmetic mean, and standard deviation were calculated. Each sample was tested three times, and the arithmetic mean, and standard deviation were computed from the results.
pH Measurement of cream formulations | Baseline
  The pH of the cosmetic emulsions was measured three times using the EcoSense® pH 10 pH/Temperature Meter, Pen Style (VMR International).
pH Measurement of cream formulations | After 12 weeks
  The pH of the cosmetic emulsions was measured three times using the EcoSense® pH 10 pH/Temperature Meter, Pen Style (VMR International).
Cream Viscosity Measurement | Baseline
  The viscosity of the cosmetic emulsions was measured three times using the RC02 rotational viscometer (Rheotec).
Light Scattering Stability Analysis | Baseline
  Stability analysis of the formulations was performed using the multiple light scattering method with the Turbiscan Lab Expert device (Formulaction SA).
Growth Factor Quantification in Cosmetic Formulations | Baseline
  The quantification of the growth factor in the obtained cosmetic formulations was conducted using a high-performance liquid chromatograph (HPLC) Varian 920-LC (Agilent Technologies), equipped with an automatic injector and sample feeder. Both qualitative and quantitative methodologies were developed for the analysis of the cosmetic preparations.
Stability Testing Points | After 2 weeks
  Stability tests for all formulations included four measurement points, analyzing the samples after 2, 4, 8, and 12 weeks of storage in climate chambers. The comprehensive testing ensured that the formulations maintained their desired properties and remained safe and effective for use throughout the study.
Stability Testing Points | After 4 weeks
  Stability tests for all formulations included four measurement points, analyzing the samples after 2, 4, 8, and 12 weeks of storage in climate chambers. The comprehensive testing ensured that the formulations maintained their desired properties and remained safe and effective for use throughout the study.
Stability Testing Points | After 8 weeks
  Stability tests for all formulations included four measurement points, analyzing the samples after 2, 4, 8, and 12 weeks of storage in climate chambers. The comprehensive testing ensured that the formulations maintained their desired properties and remained safe and effective for use throughout the study.
Stability Testing Points | After 12 weeks
  Stability tests for all formulations included four measurement points, analyzing the samples after 2, 4, 8, and 12 weeks of storage in climate chambers. The comprehensive testing ensured that the formulations maintained their desired properties and remained safe and effective for use throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Marzena Liliana Wyganowska, Prof., Study Chair — Departament of Periodontology and Oral Mucosa Diseases PUMS
Locations (1):
- Poznan University of Medical Sciences, Poznan, The Greater Poland, Poland

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and analyzed during the current study are available from the corresponding author upon reasonable request.
Supporting Information: ICF
Time Frame: 6 month after publication
Access Criteria: E-mail contact with corresponding author

REFERENCES:
- [Result] Trojahn C, Dobos G, Schario M, Ludriksone L, Blume-Peytavi U, Kottner J. Relation between skin micro-topography, roughness, and skin age. Skin Res Technol. 2015 Feb;21(1):69-75. doi: 10.1111/srt.12158. Epub 2014 Jun 3. PMID 24889351
- [Result] Dabrowska M, Mielcarek A, Nowak I. Evaluation of sex-related changes in skin topography and structure using innovative skin testing equipment. Skin Res Technol. 2018 Nov;24(4):614-620. doi: 10.1111/srt.12473. Epub 2018 Apr 29. PMID 29707820
- [Result] 12. Zalewska A., Kowalik J., Grubecki I., Application of turbiscan lab to study the effect of emulsifier content on the stability of plant origin dispersion. Chem. Process Eng. 2019; 40(4): 399-409
- [Result] Gardien KL, Baas DC, de Vet HC, Middelkoop E. Transepidermal water loss measured with the Tewameter TM300 in burn scars. Burns. 2016 Nov;42(7):1455-1462. doi: 10.1016/j.burns.2016.04.018. Epub 2016 May 24. PMID 27233677
- [Result] Dohan Ehrenfest DM, de Peppo GM, Doglioli P, Sammartino G. Slow release of growth factors and thrombospondin-1 in Choukroun's platelet-rich fibrin (PRF): a gold standard to achieve for all surgical platelet concentrates technologies. Growth Factors. 2009 Feb;27(1):63-9. doi: 10.1080/08977190802636713. PMID 19089687
- [Result] Arshdeep; Kumaran MS. Platelet-rich plasma in dermatology: boon or a bane? Indian J Dermatol Venereol Leprol. 2014 Jan-Feb;80(1):5-14. doi: 10.4103/0378-6323.125467. PMID 24448117
- [Result] Dohan Ehrenfest DM, Bielecki T, Mishra A, Borzini P, Inchingolo F, Sammartino G, Rasmusson L, Everts PA. In search of a consensus terminology in the field of platelet concentrates for surgical use: platelet-rich plasma (PRP), platelet-rich fibrin (PRF), fibrin gel polymerization and leukocytes. Curr Pharm Biotechnol. 2012 Jun;13(7):1131-7. doi: 10.2174/138920112800624328. PMID 21740379
- [Result] Feingold KR, Denda M. Regulation of permeability barrier homeostasis. Clin Dermatol. 2012 May-Jun;30(3):263-8. doi: 10.1016/j.clindermatol.2011.08.008. PMID 22507038